CLINICAL TRIAL: NCT01322555
Title: Neuroimmune Activation in Austism: Imaging Translocator Protein Using Positron Emission Tomography (PET)
Brief Title: A Study of the Association Between Autism and Immune Changes in the Brain
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110118; 11-M-0118
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-07-14

CONDITIONS: Autism Spectrum Disorders; Brain Disease; Autism; Healthy Volunteers
Keywords: PBR28; Positron Emission Tomography (PET); Propofol; Autism; Immune Response; Autism Spectrum Disorders; ASD; Healthy Volunteer; HV
MeSH Terms: conditions — Autism Spectrum Disorder; Brain Diseases; Autistic Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- People with autism and autism spectrum disorders have problems with communication, behavior, and socializing, and many also have intellectual and developmental disabilities. The cause of autism is not known, but previous research has suggested an association between autism and immune changes in the brain. Researchers are interested in using the experimental radioactive drug (11C)PBR28, which attaches to a protein in the brain that is involved in immune changes, in positron emission tomography (PET) scanning of people with and without autism to see if there are greater immune changes in those with autism.

Objectives:

- To determine if positron emission tomography scanning can be used to evaluate changes in an immune system protein in the brains of people with autism.

Eligibility:

- Individuals between 18 and 45 years of age who have been diagnosed with either autism or autism spectrum disorders, or are healthy volunteers.

Design:

* Participants will be screened with a physical examination and psychological examination, medical history, questionnaires about behavior and mood, and blood and urine tests.
* Participants will have two imaging studies of the brain at separate study visits. The first study visit will involve a magnetic resonance imaging (MRI) scan to provide a baseline image of the brain. The second study visit will involve PET scan with the radioactive chemical (11C)PBR28 to study immune system proteins in the brain. The MRI scan will take about 40 minutes, and the PET scan will take about 2 hours.
* Participants will have a final study visit 24 hours after the PET scan to provide a final blood sample for testing.

DETAILED DESCRIPTION:
Current estimates indicate that 1 in 110 children are affected with autism. Despite this striking statistic, we remain unable to describe the pathophysiology for autism, and we do not have adequate treatments for autism. The etiologies in most patients with autism are unknown, but emerging evidence supports a causal role of immune activation in autism. Multiple studies provide clear evidence of immune activation in peripheral blood of patients with autism, as demonstrated by elevations in immune markers (IFN-gamma, IL-1RA, IL-6, and TNF-alpha). Studies also demonstrate immune activation in cerebrospinal fluid (CSF) of patients with autism, as evidenced by significant elevations in cytokines and TNF-alpha. Finally, three postmortem brain studies report neuroimmune activation in patients with autism (ages 4-45). Combined, these three postmortem studies show activation of microglia and astroglia through elevations in cytokines, histology and stereology.

While the growing body of literature supporting neuroimmune activation in autism is intriguing, the current results present limitations. First, there are no studies assessing the brains of living patients with autism/ASDs. Second, the most convincing evidence for neuroimmune activation in postmortem brains is extracted almost exclusively from patients with classical autism, where intellectual disability is common. As such, the evidence for neuroimmune activation in higher functioning patients with autism and autism spectrum disorders (ASDs) is less robust.

We propose to determine whether neuroimmune activation is present in the living brains of patients with autism. Furthermore, given the heterogeneity of the autisms , as they are now called, we would like to determine whether neuroimmune activation is detectable in higher versus lower functioning patients with autism/ASDs. We propose to measure neuroimmune activation in the living brains of patients by utilizing positron emission tomography (PET) and the radioligand [(11)C]PBR28. This radioligand binds translocator protein (TSPO), which is over-expressed in activated microglia and reactive astrocytes, and has been demonstrated as a reliable marker of neuroimmune activation in various neuropsychiatric disorders. Because the majority of patients with autism/ASD will require propofol sedation to remain motionless for the two hour scan, we will include a control arm with healthy volunteers without then with propofol in order to determine the effects of propofol on [(11)C]PBR28 uptake. NIH has developed a setup in the clinical center for administering sedation/anesthesia in a safe manner, making this important study possible.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS WITH AUTISM OR ASD (INCLUSION CRITERIA):

1. Subjects must have a diagnosis of autistic disorder (299.0) or Asperger s disorder (299.80), as determined using the Diagnostic and Statistical Manual-IV (DSM-IV) and confirmation with the Autism Diagnostic Interview-Revised (Lord 1997) and/or Autism Diagnostic Observation Scale (ADOS). (A diagnosis of Pervasive Developmental Disorder, or PDD, will not suffice for this protocol).
2. Subjects must be adults between 18-45 years old.
3. Subjects must be healthy based on history and physical examination.
4. Subjects must be "binders" to [11C]PBR28 as determined via one of two ways: by prior participation in a PET scan with [11C]PBR28 or by in vitro testing of their leukocytes. We found that non-binders have markedly reduced affinity of [3H]PBR28 to leukocyte membranes. The in vitro binding has shown no overlapping values between binders (~90%) and non-binders.
5. Subjects must either provide informed consent, or they must assent in combination with informed consent by a legal guardian or durable power of attorney (DPA).

HEALTHY VOLUNTEERS (INCLUSION CRITERIA):

1. Subjects must be adults between 18-45 years old.
2. Subjects must be healthy based on history and physical examination
3. Subjects must be binders to [11 C]PBR28 (see point 4 above for details)
4. Prior to the PET scan, all healthy subjects must have had within the prior year an MRI scan of the brain to rule out significant structural abnormalities.

EXCLUSION CRITERIA:

PATIENTS WITH AUTISM OR ASD (EXCLUSION CRITERIA):

1. Any history of alcohol or substance dependence, as these conditions may alter uptake of [11C]PBR28.
2. Any history of alcohol or substance abuse within the past 6 months, as these conditions may alter uptake of [11C]PBR28.
3. Schizophrenia.
4. In addition to the diagnosis of autistic disorder, ASD or Asperger, any other Axis I disorder that requires inpatient hospitalization during this study, or is at the time of enrollment worsening relative to baseline. We will not completely exclude all Axis I disorders, because it is typical for patients with autism /ASD to carry comorbid Axis I disorders, including Generalized Anxiety Disorder (GAD), social phobia, obsessive compulsive disorder (OCD), dysthymia, Major Depressive Disorder.
5. Intellectual quotient (IQ) less than 30, as including the lowest functioning patients would make the experiment logistically challenging and would broaden heterogeneity too much.
6. Clinically significant laboratory abnormalities as assessed by the PI, medically responsible investigator or consultant.
7. Serious medical problems including but not limited to chronic neurological disease such as multiple sclerosis, autoimmune diseases, poorly controlled seizure disorder, or serious cardiopulmonary disease.
8. Active seizure disorder, as defined as having had a seizure in the past year or being on antiepileptic medications for seizures.
9. Positive HIV status.
10. Head trauma resulting in a period of unconsciousness lasting longer than 5 minutes.
11. Exposure to radiation in the past year (i.e., PET from other research), which when combined with this study would be above the allowable limits.
12. Positive urine drug screen at time of enrollment.
13. Pregnancy at time of scan (beta HCG will be measured in all female patients within 24 hours before start of scan and must be negative).
14. In patients who will get an MRI scan at NIH, metallic foreign bodies that would be affected by the MRI magnet, or a fear of enclosed spaces that would prohibit MRI scanning.
15. Allergy to propofol or eggs (since egg products are used to formulate propofol),.
16. Snoring, as this increases the likelihood of complications from propofol sedation.
17. Currently taking antibacterial drugs (such as Amoxicillin-Clavulanate/ Augmentin , Metronidazole/Flagyl Minocycline/Minocin ). We will not discontinue any medications in any subjects.
18. Currently taking antiviral drugs (such as Acyclovir/Zovirax , Interferon beta 1/Avonex , Valacyclovir/Valtrex ). We will not discontinue any medications in any subjects.
19. Taking corticosteroids within the 6 months prior to study enrollment (such as Dexamethasone/Decadron , Hydrocortisone/Hydrocortone , Methylprednisone/Medrol ). We will not discontinue any medications in any subjects.
20. Taking immunosuppressants in the past 6 months prior to study enrollment (such as Azathioprine/Imuran , Infliximab/Remicade , Sulfasalazine/ Azulfidine , Olsalazine/Dipentum ). We will not discontinue any medications in any subjects.
21. Any history of taking immunosuppressants in the context of chemotherapy or organ transplant. Medications in this class might include Tacrolimus/Prograf , 6-mercaptopurine/Purinethol , and Methotrexate/Trexall . We will not discontinue any medications in any subjects.
22. Currently taking Clozapine/Clozaril , as high doses in rats increases TSPO. With the exception of clozapine, patients may be on centrally-acting medications, including medications for mood and behavioral disturbances. These medications may be antiepileptic medications, so long as the antiepileptics are being used for symptoms of mood and behavior as opposed to seizure disorder.

Healthy Volunteers (Exclusion criteria):

1. Any past or present Axis I disorder. The exception is substance abuse which ended over 6 months prior to enrollment.
2. Intellectual disability or significant learning problems, as determined by IQ testing lower than 70, inability to read or write, or history of being unable to take regular classes while in school.
3. Clinically significant laboratory abnormalities, as defined as laboratory values that are out of normal range or require clinical workup and/or treatment.
4. With the exception of isolated doses of benzodiazepine which may be administered once or twice by the investigators of this study, psychotropic medication use (including benzodiazepines and illicit drugs) during the 28 days (42 days if fluoxetine) prior to the PET scan. Investigators of this study may administer lorazepam for anxiety (see procedures).
5. Serious medical problems including but not limited to chronic neurological disease such as multiple sclerosis, autoimmune diseases or cardiopulmonary disease that would significantly increase risk with propofol sedation.
6. Positive HIV status.
7. Metallic foreign bodies that would be affected by the MRI magnet or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
8. Head trauma resulting in a period of unconsciousness lasting longer than 5 minutes.
9. Exposure to radiation in the past year (i.e., PET from other research), which when combined with this study would be above the allowable limits.
10. Positive urine drug screen at time of enrollment
11. Inability to lie flat on a camera bed for about 2.5 hours per PET scan and 1 hour for MRI.
12. Allergy to propofol or eggs, since egg products are used to formulate propofol
13. Pregnancy at time of scan (beta HCG will be measured in all female patients within 24 hours prior to start of scan and must be negative).
14. Snoring, as this condition increases the likelihood of complications from propofol sedation.
15. Currently taking antibacterial drugs (such as Amoxicillin-Clavulanate/ Augmentin , Metronidazole/Flagyl Minocycline/Minocin ). We will not discontinue any medications in any subjects.
16. Currently taking antiviral drugs (such as Acyclovir/Zovirax , Interferon 1/Avonex , Valacyclovir/Valtrex ). We will not discontinue any medications in any subjects.
17. Taking corticosteroids within the 6 months prior to study enrollment (such as Dexamethasone/Decadron , Hydrocortisone/Hydrocortone , Methylprednisone/Medrol ). We will not discontinue any medications in any subjects.
18. Taking immunosuppressants in the past 6 months prior to study enrollment (such as Azathioprine/Imuran , Infliximab/Remicade , Sulfasalazine/ Azulfidine , Olsalazine/Dipentum ). We will not discontinue any medications in any subjects.
19. Any history of taking immunosuppressants in the context of chemotherapy or organ transplant. Medications in this class might include Tacrolimus/Prograf , 6-mercaptopurine/Purinethol , and Methotrexate/Trexall . We will not discontinue any medications in any subjects.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03-04; Study Completion 2017-07-14

PRIMARY OUTCOMES:
[11C]PBR28 uptake in brain as measured using VT (volume of distribution) and VT/fp (divided by free fraction in plasma.
Compare VT in autism versus healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baird G, Simonoff E, Pickles A, Chandler S, Loucas T, Meldrum D, Charman T. Prevalence of disorders of the autism spectrum in a population cohort of children in South Thames: the Special Needs and Autism Project (SNAP). Lancet. 2006 Jul 15;368(9531):210-5. doi: 10.1016/S0140-6736(06)69041-7. PMID 16844490
- [Background] Hertz-Picciotto I, Delwiche L. The rise in autism and the role of age at diagnosis. Epidemiology. 2009 Jan;20(1):84-90. doi: 10.1097/EDE.0b013e3181902d15. PMID 19234401
- [Background] Becker KG. Autism, asthma, inflammation, and the hygiene hypothesis. Med Hypotheses. 2007;69(4):731-40. doi: 10.1016/j.mehy.2007.02.019. Epub 2007 Apr 6. PMID 17412520
- [Derived] Paul S, Gallagher E, Liow JS, Mabins S, Henry K, Zoghbi SS, Gunn RN, Kreisl WC, Richards EM, Zanotti-Fregonara P, Morse CL, Hong J, Kowalski A, Pike VW, Innis RB, Fujita M. Building a database for brain 18 kDa translocator protein imaged using [11C]PBR28 in healthy subjects. J Cereb Blood Flow Metab. 2019 Jun;39(6):1138-1147. doi: 10.1177/0271678X18771250. Epub 2018 May 11. PMID 29749279